STUDY TITLE: A Pilot Feasibility Study of Mindfulness-Oriented Recovery Enhancement with Pregnant Women with Opioid Use Disorder

Clinicaltrials.gov Identifier: NCT04824521

PRINCIPAL INVESTIGATOR: Sarah Reese, School of Social Work, University of Montana, 406-243-

5543

DOCUMENT DATE: February 10, 2021

ATTACHMENTS:

Statistical Analysis Plan

## Statistical Analysis Plan

I will calculate means and standard deviations for all self-report measures. I will analyze the data Semi-structured interview recordings will be transcribed verbatim by a professional transcription company, Rev.com. Along with two trained research assistants, I will follow Braun and Clarke's six-phase approach to thematic data analysis. <sup>64</sup> First, becoming familiar with the data, then generating initial codes, searching for themes, reviewing themes, defining and naming themes, and finally, producing a report. We will use NVivo software to organize data when coding transcripts.